CLINICAL TRIAL: NCT03056001
Title: A Pilot Study Evaluating the Safety, Tolerability, and Efficacy of Doxorubicin and Pembrolizumab in Patients With Metastatic or Unresectable Soft Tissue Sarcoma
Brief Title: Safety, Tolerability, and Efficacy of Doxorubicin and Pembrolizumab for Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081342; 00020377; LCI-SAR-STS-PEM-001 (Other: Atrium Health)
Record Dates: First submitted 2017-02-03; First posted 2017-02-16 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Soft Tissue Sarcoma, Adult; Soft Tissue Sarcoma, Child
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + doxorubicin (Experimental): Participants will receive pembrolizumab IV infusion and doxorubicin IV injection on Day 1 of every 21 (+/- 3) days
  Interventions: Drug: Pembrolizumab; Drug: Doxorubicin

INTERVENTIONS:
Drug: Pembrolizumab — IV infusion on day 1 of each 3 week cycle, at dose of 200 mg
  Other Names: KEYTRUDA®
Drug: Doxorubicin — IV injection on day 1 of each 3 week cycle, starting at dose of 60 mg/m2 (may be escalated to 75 mg/m2 per investigator discretion after Cycle 1)
  Other Names: Adriamycin

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of doxorubicin in combination with pembrolizumab in subjects with metastatic or unresectable soft tissue sarcoma. Based on previous studies, pembrolizumab may be an effective study treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and toxicity profile of doxorubicin and pembrolizumab in previously treated or untreated subjects with unresectable or metastatic soft tissue sarcoma. The secondary objectives are to assess overall survival, and response rate, duration of response, and progression-free survival (PFS) with this regimen using RECIST 1.1 criteria. The exploratory objectives are to assess PFS, overall response rate, duration of response, and disease control rate using the immune-related RECIST (irRECIST) criteria, evaluate the correlation between PD-L1 expression levels and antitumor activity of MK-3475, investigate other biomarkers that may correlate with tumor responses, and evaluate differences in tumor tissue characteristics in biopsies taken during or post-treatment with MK-3475 versus baseline.

ELIGIBILITY:
Inclusion Criteria

1. Be willing and able to provide written informed consent for the trial.
2. Must have a histologically confirmed diagnosis of unresectable or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy. Patients with Ewings sarcoma, osteosarcoma, chondrosarcoma, Kaposis sarcoma, gastrointestinal stromal tumors (GIST), clear cell sarcoma, alveolar soft part sarcoma and any other soft tissue or bone sarcoma felt to be chemotherapy resistant in the opinion of the Sponsor-Investigator will be excluded.
3. Must not have received prior treatment with an anthracycline chemotherapy (eg, doxorubicin) and/or anti-PD-1/PD-L1 therapy.
4. May have had any number of prior systemic cytotoxic therapies for unresectable/metastatic disease.
5. Must have at least one radiologically measurable lesion as per RECIST 1.1 defined as a lesion that is 10mm in longest diameter or lymph node that is 15mm in short axis imaged by CT scan or MRI. Tumors with previously irradiated field will be designated as nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence of at least 90 days following completion of radiotherapy.
6. All subjects with accessible tumor will be asked to provide a fresh tumor biopsy if they can be safely biopsied in the opinion of the investigator. Recently obtained archived core or excisional biopsy of a tumor lesion (obtained up to 12 months prior to Cycle 1 Day 1) may be substituted only if the subject is unwilling or unable (e.g. inaccessible or subject safety concern) to undergo a fresh tumor biopsy. Subjects who are unwilling or unable to have a fresh tumor biopsy and do not have recently obtained archived tissue available may submit an archived specimen (obtained > 12 months prior to Cycle 1 Day 1) only upon approval from the Sponsor-Investigator.
7. Be at least 12 years of age on day of signing informed consent. Assent will be obtained in appropriately aged subjects per institutional guidelines.
8. ECOG performance status 0 or 1.
9. Life expectancy of at least 3 months per the Investigator.
10. Have adequate organ function as indicated by the laboratory values in Table 1 of protocol. All screening labs should be performed within 10 days of treatment initiation. PT/INR and PTT must be performed within 7 days of study treatment initiation for subjects on anti-coagulants such as coumadin/heparin.
11. The subject has left ventricular ejection fraction (LVEF) greater than or equal to 50% assessed within 21 days prior to study regimen initiation.
12. Subjects must not be expecting to conceive or father children within the timeframe referenced below. Subjects of childbearing potential must be willing to adhere to the contraception requirement as described in Section 3.3.2 from the day of the screening visit (or 14 days prior to the initiation of study treatment for oral contraception) throughout the study period up to 120 days after the last dose of pembrolizumab and/or up to 180 days after the last dose of doxorubicin. If there is any question that a subject of childbearing potential will not reliably comply with the requirements for contraception, that subject should not be entered into the study.
13. Female subjects of childbearing potential must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study treatment). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the subject to be eligible.
14. Subject has voluntarily agreed to participate by giving written informed consent for the trial. The subject may also provide consent for Optional and Future Studies-Biospecimen Collection. However, the subject may participate in the main trial without participating in Optional and Future Studies.

Exclusion Criteria

1. Currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 30 days of the first dose of study regimen.
2. Have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study regimen.
3. Have a known history of active TB (Bacillus Tuberculosis).
4. Have had a prior anti-cancer monoclonal antibody (mAb) given to treat malignancy within 4 weeks prior to the first dose of study regimen or have not recovered (i.e. less than or equal to Grade 1 or at baseline) from adverse events due to previous mAbs.
5. Have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of study regimen or who have not recovered (i.e. less than or equal to Grade 1 or at baseline) from adverse events due to previous chemotherapy, targeted small molecule therapy, or radiation therapy.

   Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

   Note: If subjects have received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy as determined by the Investigator.
6. Have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
7. Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study regimen and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to the first dose of the study regimen. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
8. Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Have known history of, or any evidence of active, non-infectious pneumonitis.
10. Have an active infection requiring systemic therapy (uncomplicated urinary tract infection treated with oral antibiotics is permitted).
11. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects participation for the full duration of the trial, or is not in the best interest of the subjects to participate, in the opinion of the treating Investigator.
12. Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as determined by the Investigator.
13. Are pregnant or breastfeeding
14. Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Have a known history of Human Immunodeficiency Virus infection (e.g. HIV 1/2 antibodies).
16. Have known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA [qualitative] is detected).
17. Have received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Jagosky, MD, Principal Investigator — Levine Cancer Institute, Atrium Health (formerly Carolinas HealthCare System)
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Search clinical trials at Levine Cancer Institute. — https://www.carolinashealthcare.org/research-clinical-trials/cancer-clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Doxorubicin
Started | 30
Completed | 6
Not Completed | 24
Not completed — Death | 24

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 61.5 [21 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 23
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 30
Primary Tumor Site [Count of Participants; unit: Participants]
  Extremity - Arm | 2
  Extremity - Leg | 8
  Retroperitoneal/Abdomen | 13
  Other | 7
Histology [Count of Participants; unit: Participants]
  Liposarcoma | 7
  Leiomyosarcoma | 10
  Synovial Sarcoma | 1
  Undifferentiated Pleomorphic Sarcoma | 4
  Angiosarcoma | 2
  Rhabdomyosarcoma | 1
  Epithelioid angiosarcoma | 1
  Fibromyxoid sarcoma/sclerosing epithelioid fibrosarcoma | 1
  Malignant fibrous histiocytoma | 1
  Spindle cell solitary fibrous tumor | 1
  Extraskeletal osteosarcoma | 1
Metastatic Site [Count of Participants; unit: Participants]
  Liver | 6
  Lung | 8
  Lymph Node | 2
  Other | 13
  N/A - no metastatic disease | 1
Prior Lines of Systemic Treatment for Sarcoma [Count of Participants; unit: Participants]
  0 prior lines | 25
  1 prior line | 2
  2 prior lines | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Severe or Life-Threatening Adverse Event
Description: Severe or life-threatening adverse events will be determined for each subject as a binary variable indicating whether or not the subject experienced at least one adverse event that meets the following criteria: is considered a serious adverse event (per CFR 21 Part 312), is study treatment related per the Sponsor-Investigator, and considered to be clinically significant by the Sponsor-Investigator. An adverse event will be considered study treatment related if it is determined that the event is at least possibly related to either pembrolizumab, doxorubicin, or both.
Time Frame: From enrollment to at least 90 days following cessation of study treatment. The median time on treatment was 5.8 months.
Population: The evaluable population will consist of all subjects who begin study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 30
Participants | 1
Statistical Analysis 1: Comparison: Pembrolizumab + Doxorubicin; The reported severe or life-threatening adverse event rate with weekly doxorubicin and dacarbazine was 0.55. If it became evident that the rate of severe or life-threatening toxicity convincingly exceeded 0.55, the study would have been halted. Convincing evidence of exceeding 0.55 was based on Bayesian methods and continuous monitoring, where the stopping rule would have held enrollment if the posterior probability at any point exceeded 0.75 or higher; Test type: Other — Estimation only; Rate = 0.0333, 95% CI 2-sided [0.0008 to 0.1722] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from treatment start date to the date of death from any cause. Subjects who are alive or lost to follow up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From treatment start to date of death, or censored as described; assessed for approximately 5 yrs or until censoring rate for entire study reduced to 20%, whichever occurred first. When the censoring rate reached 20%, OS time ranged from 0.1 - 4.8 yrs.
Population: The evaluable population consisted of all enrolled subjects who began study therapy.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 30
years | 1.3 [0.8 to 2.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Doxorubicin; Test type: Other — Estimation only; Median = 1.3, 95% CI 2-sided [0.8 to 2.1] — The Kaplan Meier method was used to estimate the median OS (in years) for the population. The Greenwood method was used to estimate the confidence limits of the median overall survival

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from enrollment to time of progression or death. Disease progression (PD) may be determined objectively per RECIST 1.1 (Response Evaluation Criteria in Solid Tumors, where PD is defined as a 20% increase in the sum of longest diameters of target lesions, a measurable increase in non-target lesion, or appearance of new lesions) or subjectively as determined by investigator (with evidence documented in the medical records). If the subject died without documented PD, date of progression will be date of death. For surviving subjects who did not have documented PD, PFS was censored at last radiologic assessment. For subjects who received subsequent anticancer therapy prior to documented PD, PFS was censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who experienced a PFS event following an interval equal to two or more scheduled radiologic assessments were censored at last assessment prior to first missed assessment.
Time Frame: From treatment start date to date of progression/death, or censored as described; assessed for approximately 2 years.
Population: The evaluable population consisted of all enrolled subjects who began study therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 30
months | 5.7 [4.1 to 8.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Doxorubicin; Test type: Other — Estimation only; Median = 5.7, 95% CI 2-sided [4.1 to 8.3] — The Kaplan Meier method was used to estimate the median PFS (in months) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival

4. Secondary Outcome: Number of Subjects With an Objective Response
Description: Objective response was determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR) or partial response (PR) as determined by RECIST 1.1 response criteria. A CR is indicated by disappearance of all target and non target lesions. A PR is indicated by >=30% decrease in sum of longest diameter of target lesions with baseline as reference.
Time Frame: From enrollment to best response while on study treatment; subjects remained on treatment until disease progression or death or unacceptable toxicity (subjects were on treatment for a median of 5.8 months)
Population: The evaluable population will consist of all subjects who begin study therapy and have measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 30
Participants | 11
Statistical Analysis 1: Comparison: Pembrolizumab + Doxorubicin; Test type: Other — Estimation only; Rate = 0.367, 95% CI 2-sided [0.199 to 0.561] — Confidence interval estimated using the Clopper Pearson method

5. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) is defined as the duration of time from the first assessment that determined a CR or PR to the date of the first occurrence of progressive disease or death. Progression events and the censoring mechanism for DoR will be the same as described for PFS. DoR will be determined for each subject using the RECIST 1.1 criteria.
Time Frame: From date of response to date of progression/death, or censored as described above; assessed for approximately 2 years.
Population: The evaluable population consisted of all enrolled subjects who begin study therapy and achieve objective response (CR or PR) on study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab + Doxorubicin
Number analyzed (Participants) | 11
months | 8.0 [2.8 to 34.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Doxorubicin; Test type: Other — Estimation only; Median = 8.0, 95% CI 2-sided [2.8 to 34.6] — The Kaplan Meier method was used to estimate the median DoR (in months) for the population. The Greenwood method was used to estimate the confidence limits of the median duration of response

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and through 30 days after last dose of study treatment, an average of 7.3 months.
Arm/Group | Pembrolizumab + Doxorubicin
All-Cause Mortality (participants affected / at risk) | 24/30
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Doxorubicin (N=30)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Adrenal insufficiency (Endocrine disorders) | 1 — Hypophysitis
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Death NOS (General disorders) | 2
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Failure to thrive
Cholecystitis (Hepatobiliary disorders) | 1
Autoimmune disorder (Immune system disorders) | 1 — Hepatitis
Infections and infestations - Other, specify (Infections and infestations) | 1 — Bacteremia
Lung infection (Infections and infestations) | 3 — Pneumonia
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Doxorubicin (N=30)
Anemia (Blood and lymphatic system disorders) | 10
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — varicosites
Leukocytosis (Blood and lymphatic system disorders) | 1
Spleen disorder (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 — cold intolerance
Endocrine disorders - Other, specify (Endocrine disorders) | 1 — low testosterone
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — altered vision
Watering eyes (Eye disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Tongue Discoloration
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 22
Oral pain (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 2
Rectal perforation (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Chills (General disorders) | 6
Edema face (General disorders) | 2
Edema limbs (General disorders) | 3
Facial pain (General disorders) | 1
Fatigue (General disorders) | 19
Fever (General disorders) | 7
Flu like symptoms (General disorders) | 1
Gait disturbance (General disorders) | 1
Localized edema (General disorders) | 3
Malaise (General disorders) | 5
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 — Yeast Infection
Infections and infestations - Other, specify (Infections and infestations) | 1 — Shingles left butt
Lung infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 5
Ejection fraction decreased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1 — ACTH level low
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 4
Serum amylase increased (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — hand tenderness
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — jaw pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — swelling of hand
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Sebaceous cysts
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 5
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Pyuria
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 2
Urine discoloration (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Obstructive airway
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — scattered rhonchi
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Erythema R Buttock
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — nail discomfort
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — sun damage on chest
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Petechia
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — lip sores
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — facial erythema
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Erythema- Cellulitis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — skin ulceration port site
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Thromboembolic event (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT03056001/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03056001/ICF_001.pdf